CLINICAL TRIAL: NCT00906347
Title: A Randomized, Controlled Trial of Oral Misoprostol for Labor Augmentation
Brief Title: A Trial of Oral Misoprostol for Labor Augmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102008-030
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2009-05

CONDITIONS: Labor Augmentation
Keywords: Labor augmentation; Oral misoprostol
MeSH Terms: interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin augmentation (Active Comparator): Women with hypotonic labor and a clinical decision to proceed with labor augmentation will receive intravenous oxytocin.
  Interventions: Drug: Oxytocin
- Misoprostol augmentation (Active Comparator): Women with hypotonic labor and a clinical decision to proceed with labor augmentation will receive oral misoprostol.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 75 micrograms orally every 4 hours for up to 2 doses.
  Other Names: Cytotec
  Arms: Misoprostol augmentation
Drug: Oxytocin — Intravenous oxytocin will be administered per the established Labor and Delivery protocol at Parkland Memorial Hospital
  Other Names: Pitocin
  Arms: Oxytocin augmentation

SUMMARY:
This is a prospective, randomized, controlled trial designed to examine the efficacy of oral misoprostol for labor augmentation compared to a standard regimen of intravenous oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* Clinical decision to augment labor
* Gestational age > than or equal to 36 weeks
* Singleton gestation
* Cephalic presentation
* Reassuring fetal heart rate tracing
* Cervical dilation between 4 and 8 cm
* Ruptured membranes with clear amniotic fluid
* Intrauterine pressure catheter in place
* Less than 200 MVUs in a 10 minute period
* 5 or fewer contractions in a 10 minute period
* English or Spanish speaking patient

Exclusion Criteria:

* Non-reassuring fetal heart rate tracing at time of enrollment
* Meconium stained amniotic fluid
* Previous uterine incision
* Maternal fever (defined as greater than 37.9 C)
* Known fetal anomalies
* Placenta previa or unexplained vaginal bleeding
* Estimated fetal weight of 4,500 grams or more
* Abnormal maternal bony pelvis
* Grandmultiparity

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: April Bleich, MD, Principal Investigator — University of Texas Southwestern Medical Center; Kenneth Leveno, MD, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Bleich AT, Villano KS, Lo JY, Alexander JM, McIntire DD, Leveno KJ. Oral misoprostol for labor augmentation: a randomized controlled trial. Obstet Gynecol. 2011 Dec;118(6):1255-1260. doi: 10.1097/AOG.0b013e318236df5b. PMID 22105254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women presenting to Labor and Delivery at Parkland Memorial Hosiptal and who met eligibility requirements were offered participation from Decemeber 2008 through January 2001.
Groups:
- Misoprostol Augmentation: Women with hypotonic labor and a clinical decision to proceed with labor augmentation will receive oral misoprostol.
  Misoprostol : 75 micrograms orally every 4 hours for up to 2 doses.
- Oxytocin Augmentation: Women with hypotonic labor and a clinical decision to proceed with labor augmentation will receive intravenous oxytocin.
  Oxytocin : Intravenous oxytocin will be administered per the established Labor and Delivery protocol at Parkland Memorial Hospital
Period: Randomized
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Started | 176 | 174
Completed | 176 | 174
Not Completed | 0 | 0
Period: Received Study Drug
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Started | 176 | 174
Completed | 136 | 143
Not Completed | 40 | 31
Not completed — 8 cm prior to initiation of study drug | 18 | 30
Not completed — Nonreassuring fetal heart rate | 13 | 1
Not completed — Refused study drug | 1 | 0
Not completed — Uterine tachysystole or hypertonus | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation | Total
Number analyzed (Participants) | 176 | 174 | 350
Age, Customized [Mean (Standard Deviation); unit: years] | 24.9 (5.8) | 24.1 (5.3) | 24.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 174 | 350
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 176 | 174 | 350

OUTCOME MEASURES:

1. Primary Outcome: Uterine Tachysystole
Description: Defined as six contractions in two consecutive 10-minute periods
Time Frame: Up to four hours after administration of study drug
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Number analyzed (Participants) | 176 | 174
participants | 50 | 41

2. Secondary Outcome: Infant Apgar Score <4
Description: Assigned on a scale of 0-10 by pediatric provider attending delivery. A lower score reflects need for further resuscitation and is potentially associated with increased risk of adverse neurological outcomes.
Time Frame: 5 minutes after delivery
Population: Intent to treat
Measure: Number; unit: infants
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Number analyzed (Participants) | 176 | 174
infants | 0 | 0

3. Secondary Outcome: Umbilical Cord Artery pH <7.1
Time Frame: Obtained at delivery
Population: Intent to treat
Measure: Number; unit: infants
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Number analyzed (Participants) | 176 | 174
infants | 3 | 4

4. Secondary Outcome: Admission of Neonatal Intensive Care Unit
Time Frame: Until hospital discharge
Population: Intent to treat
Measure: Number; unit: infants
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Number analyzed (Participants) | 176 | 174
infants | 1 | 0

5. Secondary Outcome: Maternal Chorioamnionitis
Description: Temperature 38 degrees C or higher in the absence of other sources of infection
Time Frame: During labor
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Number analyzed (Participants) | 176 | 174
participants | 28 | 32

6. Secondary Outcome: Maternal Hypovolemia Requiring Blood Transfusion
Time Frame: Until hospital discharge
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Number analyzed (Participants) | 176 | 174
participants | 6 | 2

7. Secondary Outcome: Method of Delivery
Time Frame: At delivery
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Number analyzed (Participants) | 176 | 174
participants
  Spontaneous vaginal | 153 | 154
  Forceps | 4 | 2
  Cesarean for dystocia | 11 | 13
  Cesarean for nonreassuring fetal heart rate | 8 | 5

8. Secondary Outcome: Time Elapsed From Start of Labor Augmentation to Delivery
Time Frame: Initiation of augmentation until delivery
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Number analyzed (Participants) | 176 | 174
minutes | 306 [150 to 534] | 276 [162 to 462]

ADVERSE EVENTS:
Time Frame: During study period
Arm/Group | Misoprostol Augmentation | Oxytocin Augmentation
Serious Adverse Events (participants affected / at risk) | 1/176 | 2/174
Other Adverse Events (participants affected / at risk) | 0/176 | 0/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misoprostol Augmentation (N=176) | Oxytocin Augmentation (N=174)
Need for emergent cesarean delivery secondary to nonreassuirng fetal heart rate (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No